CLINICAL TRIAL: NCT02080715
Title: A Randomized, Double-blind, Placebo-controlled Examination of the Effects of Tolcapone (TASMAR) on Vigilance in Healthy Volunteers After Sleep Deprivation
Brief Title: Role of the Catechol-O-methyltransferase (COMT) in the Physiological Regulation of Vigilance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: COMT and vigilance
Record Dates: First submitted 2013-10-10; First posted 2014-03-06 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Sleep-wake; regulation; volunteers
MeSH Terms: interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolcapone (Experimental): Tasmar
  Interventions: Drug: Tolcapone; Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — 2 x 100mg Tolcapone compared to placebo (randomized, double-blind, cross-over)
  Other Names: Tasmar
Drug: Placebo

SUMMARY:
In this study, pharmacologic effects of COMT inhibition during sleep deprivation in healthy subjects in dependence of their Val158Met genotype of COMT are studied. Potential effects are identified by measurement of vigilance and cognitive performance as well as EEG measurements during wake and sleep.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects
* Age: 20-30 years
* written informed consent
* right handed
* non smoker

Exclusion criteria:

* sleep disturbances
* irregular sleep-wake rhythm
* travelling with time-shift
* liver diseases (ALT: > 82 U/l; AST: > 76 U/l)
* diseases of the nervous system
* acute internal medicine diseases
* medication or drug abuse
* intake of more than 3 caffeine-containing drinks
* intake of more than 5 alcoholic drinks per week
* heart pacemaker or implanted medical devices
* Body-Mass-Index (BMI): 20< BMI >26

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evolution of vigilance during prolonged wakefulness after intake of tolcapone when compared to placebo | Participants will be studied during two weeks
  Vigilance is measured subjectively (questionnaires and visual analogue scales) and objectively (e.g., psychomotor vigilance task: reaction times and number of lapses; waking EEG: spectral power) at 3-hour intervals during 40 hours prolonged wakefulness in 30 healthy male adults.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Landolt, Professor, Study Chair — University of Zurich, Institute of Pharmacology and Toxicology; Christian Baumann, MD, Principal Investigator — University Hospital Zurich, Department of Neurology
Locations (1):
- University of Zurich, Institute of Pharmacology and Toxicology, Zurich, Switzerland